CLINICAL TRIAL: NCT06041087
Title: Dairy Supplementation and the Post-Exercise Bone and Inflammatory Response
Brief Title: Bone and Inflammatory Outcomes - Nutrition and Exercise Trials
Acronym: BIONEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Andrea Josse, Assistant Professor, York University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-045b
Record Dates: First submitted 2023-08-25; First posted 2023-09-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Bone; Inflammation
Keywords: Bone health; Females; Dairy; Exercise; Inflammation
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — High-Intensity Interval Training; Carbohydrates; Water; Milk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise and Greek Yogurt (GY) (Experimental): Participants will have a fasted baseline blood sample taken upon arrival to the lab. Then they will take part in a high-intensity exercise protocol, consisting of high-intensity interval cycling, resistance exercise, and plyometrics. Following exercise, participants will return to the lab for a 5min post-exercise blood sample, and then consume ~200g Greek yogurt (0% milk fat). An additional blood sample will be taken at 1h post-exercise, followed by an additional ~200g of Greek yogurt. Blood samples will also be taken at 4h and 24h post-exercise. Participants will also rate their muscle soreness and perform a jump height test at pre-exercise, 5min post-exercise, 4h and 24h post-exercise.
  Interventions: Behavioral: High-Intensity Exercise; Dietary Supplement: Greek yogurt
- Exercise and Milk (Milk) (Experimental): Participants will have a fasted baseline blood sample taken upon arrival to the lab. Then they will take part in a high-intensity exercise protocol, consisting of high-intensity interval cycling, resistance exercise, and plyometrics. Following exercise, participants will return to the lab for a 5min post-exercise blood sample, and then consume ~500ml plain skim milk (0% milk fat). An additional blood sample will be taken at 1h post-exercise, followed by an additional ~500ml of skim milk. Blood samples will also be taken at 4h and 24h post-exercise. Participants will also rate their muscle soreness and perform a jump height test at pre-exercise, 5min post-exercise, 4h and 24h post-exercise.
  Interventions: Behavioral: High-Intensity Exercise; Dietary Supplement: Skim Milk
- Exercise and Carbohydrate (CHO) (Active Comparator): Participants will have a fasted baseline blood sample taken upon arrival to the lab. Then they will take part in a high-intensity exercise protocol, consisting of high-intensity interval cycling, resistance exercise, and plyometrics. Following exercise, participants will return to the lab for a 5min post-exercise blood sample, and then consume ~50g of maltodextrin mixed with water (~500ml). An additional blood sample will be taken at 1h post-exercise, followed by an additional ~500ml of the maltodextrin drink. Blood samples will also be taken at 4h and 24h post-exercise. Participants will also rate their muscle soreness and perform a jump height test at pre-exercise, 5min post-exercise, 4h and 24h post-exercise.
  Interventions: Behavioral: High-Intensity Exercise; Dietary Supplement: Carbohydrate (Maltodextrin powder mixed with water)
- Exercise and Water (W) (Placebo Comparator): Participants will have a fasted baseline blood sample taken upon arrival to the lab. Then they will take part in a high-intensity exercise protocol, consisting of high-intensity interval cycling, resistance exercise, and plyometrics. Following exercise, participants will return to the lab for a 5min post-exercise blood sample, and then consume ~500ml water. An additional blood sample will be taken at 1h post-exercise, followed by an additional ~500ml water. Blood samples will also be taken at 4h and 24h post-exercise. Participants will also rate their muscle soreness and perform a jump height test at pre-exercise, 5min post-exercise, 4h and 24h post-exercise.
  Interventions: Behavioral: High-Intensity Exercise; Dietary Supplement: Water

INTERVENTIONS:
Behavioral: High-Intensity Exercise — A single bout of high-intensity exercise (cycling intervals, resistance exercise, plyometrics) per trial.
Dietary Supplement: Carbohydrate (Maltodextrin powder mixed with water) — 50g consumed immediately after exercise and 1h after exercise.
  Other Names: CHO
  Arms: Exercise and Carbohydrate (CHO)
Dietary Supplement: Skim Milk — 500ml consumed immediately after exercise and 1h after exercise.
  Other Names: Milk
  Arms: Exercise and Milk (Milk)
Dietary Supplement: Greek yogurt — 200g consumed immediately after exercise and 1h after exercise.
  Other Names: GY
  Arms: Exercise and Greek Yogurt (GY)
Dietary Supplement: Water — 500ml consumed immediately after exercise and 1h after exercise.
  Other Names: W
  Arms: Exercise and Water (W)

SUMMARY:
This study investigates whether dairy products will positively impact loading exercise-induced bone turnover and bone cell activity and/or the post-exercise inflammatory response in healthy young adults compared to a carbohydrate drink and/or water.

DETAILED DESCRIPTION:
Introduction: Two million individuals at a cost of around 4.6 billion dollars a year in Canada suffer from osteoporosis. It is important to investigate strategies that can reduce bone loss and/or increase bone mass. Similarly, inflammation is associated with many different disease states, and investigating strategies to reduce systemic inflammation is prudent. Nutrition and exercise may be inexpensive and accessible strategies to improve bone health and inflammation and should be explored in different contexts and implemented. Our proposed research combines both nutrition and exercise along with the assessment of bone turnover and inflammatory markers in healthy young adults.

Design: Randomized controlled crossover trial

Participants: Healthy, university aged males and females.

Methods: During the study participants will complete 4 different acute exercise and nutritional supplement trials, in random order. The four trials are: 1) exercise+carbohydrate (CHO), 2) exercise+milk (Milk), 3) exercise+Greek yogurt (GY), and 4) exercise+water (W). The whole study will take a maximum of 16 weeks and each supplement trial will be separated by 2-4 weeks.

Outcomes: several markers of bone turnover and bone cell activity as well as markers of inflammation will be measured in the blood, before exercise and at different times post-exercise and post supplement consumption.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years
* Normal BMI (18.5-24.9) kg/m^2
* Low to moderately physically active (0-2 times/week)
* No allergy to dairy protein or lactose intolerance
* On no medication related to a chronic condition
* On birth control or naturally cycling with a regular menstrual cycle)

Exclusion Criteria:

* Regular smoker (cigarettes, e-cigarettes (e.g., vapes) or cannabis)
* Any chronic condition, inflammatory, or auto-immune condition

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Acute Bone Turnover/Cell Activity | Pre-exercise
  OPG measured in serum/plasma
Acute Bone Turnover/Cell Activity | Pre-exercise
  RANKL measured in serum/plasma
Acute Bone Turnover/Cell Activity | Pre-exercise
  OC measured in serum/plasma
Acute Bone Turnover/Cell Activity | Pre-exercise
  SOST measured in serum/plasma
Acute Bone Turnover/Cell Activity | Pre-exercise
  CTX measured in serum/plasma
Acute Bone Turnover/Cell Activity | 5 minutes post-exercise
  OPG measured in serum/plasma
Acute Bone Turnover/Cell Activity | 5 minutes post-exercise
  RANKL measured in serum/plasma
Acute Bone Turnover/Cell Activity | 5 minutes post-exercise
  OC measured in serum/plasma
Acute Bone Turnover/Cell Activity | 5 minutes post-exercise
  SOST measured in serum/plasma
Acute Bone Turnover/Cell Activity | 5 minutes post-exercise
  CTX measured in serum/plasma
Acute Bone Turnover/Cell Activity | 1 hour post-exercise
  OPG measured in serum/plasma
Acute Bone Turnover/Cell Activity | 1 hour post-exercise
  RANKL measured in serum/plasma
Acute Bone Turnover/Cell Activity | 1 hour post-exercise
  OC measured in serum/plasma
Acute Bone Turnover/Cell Activity | 1 hour post-exercise
  SOST measured in serum/plasma
Acute Bone Turnover/Cell Activity | 1 hour post-exercise
  CTX measured in serum/plasma
Acute Bone Turnover/Cell Activity | 4 hours post-exercise
  OPG measured in serum/plasma
Acute Bone Turnover/Cell Activity | 4 hours post-exercise
  RANKL measured in serum/plasma
Acute Bone Turnover/Cell Activity | 4 hours post-exercise
  OC measured in serum/plasma
Acute Bone Turnover/Cell Activity | 4 hours post-exercise
  SOST measured in serum/plasma
Acute Bone Turnover/Cell Activity | 4 hours post-exercise
  CTX measured in serum/plasma
Acute Bone Turnover/Cell Activity | 24 hours post-exercise
  OPG measured in serum/plasma
Acute Bone Turnover/Cell Activity | 24 hours post-exercise
  RANKL measured in serum/plasma
Acute Bone Turnover/Cell Activity | 24 hours post-exercise
  OC measured in serum/plasma
Acute Bone Turnover/Cell Activity | 24 hours post-exercise
  SOST measured in serum/plasma
Acute Bone Turnover/Cell Activity | 24 hours post-exercise
  CTX measured in serum/plasma
Systemic Inflammation - Serum/Plasma Cytokines | Pre-exercise
  TNF-alpha measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | Pre-exercise
  IL-6 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | Pre-exercise
  IL-1B measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | Pre-exercise
  IL-10 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 5 minutes post-exercise
  TNF-alpha measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 5 minutes post-exercise
  IL-6 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 5 minutes post-exercise
  IL-1B measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 5 minutes post-exercise
  IL-10 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 1 hour post-exercise
  TNF-alpha measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 1 hour post-exercise
  IL-6 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 1 hour post-exercise
  IL-1B measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 1 hour post-exercise
  IL-10 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 4 hours post-exercise
  TNF-alpha measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 4 hours post-exercise
  IL-6 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 4 hours post-exercise
  IL-1B measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 4 hours post-exercise
  IL-10 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 24 hours post-exercise
  TNF-alpha measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 24 hours post-exercise
  IL-6 measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 24 hours post-exercise
  IL-1B measured in serum/plasma.
Systemic Inflammation - Serum/Plasma Cytokines | 24 hours post-exercise
  IL-10 measured in serum/plasma.
Systemic inflammation - Immune Cells | Pre-exercise
  Leukocytes measured via flow cytometry
Systemic inflammation - Immune Cells | 1 hour post-exercise
  Leukocytes measured via flow cytometry
Systemic inflammation - Immune Cells | 4 hours post-exercise
  Leukocytes measured via flow cytometry
Systemic inflammation - Immune Cells | 24 hours post-exercise
  Leukocytes measured via flow cytometry

SECONDARY OUTCOMES:
Muscle soreness | Pre-exercise
  Muscle soreness rated on a 0-5 scale.
Muscle soreness | 5 minutes post-exercise
  Muscle soreness rated on a 0-5 scale.
Muscle soreness | 4 hours post-exercise
  Muscle soreness rated on a 0-5 scale.
Muscle soreness | 24 hours post-exercise
  Muscle soreness rated on a 0-5 scale.
Performance - Jump Height | Pre-exercise
  Vertical jump height measured using a counter movement jump technique.
Performance - Jump Height | 5 minutes post-exercise
  Vertical jump height measured using a counter movement jump technique.
Performance - Jump Height | 4 hours post-exercise
  Vertical jump height measured using a counter movement jump technique.
Performance - Jump Height | 24 hours post-exercise
  Vertical jump height measured using a counter movement jump technique.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Josse, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No